CLINICAL TRIAL: NCT02879682
Title: Randomized Controlled Multicenter Trial on the Impact of Presurgical Navigated Transcranial Magnetic Stimulation for Motor Mapping of Rolandic Lesions
Brief Title: nTMS for Motor Mapping of Rolandic Lesions
Acronym: Motorstim
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Charite University, Berlin, Germany (Other); Evangelisches Krankenhaus Bielefeld gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 5496/12
Record Dates: First submitted 2016-08-12; First posted 2016-08-26 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Glioma; Brain Metastases
Keywords: glioma; brain metastases; nTMS
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: preoperative Mapping
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nTMS (Active Comparator): presurgical motor mapping by nTMS and fusion with intraoperative neuronavigation
  Interventions: Procedure: nTMS data available for the surgeon
- non-nTMS (Sham Comparator): presurgical motor mapping by nTMS without access of the surgeon to these data
  Interventions: Procedure: nTMS data not available for the surgeon

INTERVENTIONS:
Procedure: nTMS data available for the surgeon — the preoperatively acquired map of the motor cortex by nTMS will be available for the surgeon
  Arms: nTMS
Procedure: nTMS data not available for the surgeon — the preoperatively acquired map of the motor cortex by nTMS will not be available for the surgeon
  Arms: non-nTMS

SUMMARY:
To compare presurgical motor mapping by navigated transcranial magnetic stimulation for surgery (nTMS) of rolandic lesions to surgery with mapping without implementing these data into neuronavigation as control.

Primary objective: Permanently new postoperative deficit is lower when the preoperative motor mapping is available to the surgeon

DETAILED DESCRIPTION:
Experimental intervention:

presurgical motor mapping by navigated transcranial magnetic stimulation and fusion with intraoperative neuronavigation

Control intervention:

presurgical motor mapping by navigated transcranial magnetic stimulation without access of the surgeon to this data Follow-up per patient: 6 months Duration of intervention per patient: 45 minutes

ELIGIBILITY:
Key inclusion criteria:

* indication for resection of a supratentorial tumor within or adjacent to the primary motor cortex
* preoperative nTMS mapping of the ipsilateral hemisphere
* implementation of the mapping data into preoperative planning
* continuous MEP monitoring - informed consent

Key exclusion criteria:

* no motor eloquent tumor
* infratentorial tumor
* no postoperative imaging
* prognosis lower than 3 months of survival - age <18 years

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Operation-related neurological motor deficit 3 months after surgery as measured by NIHSS scale | 3 months after surgery
  deterioration in NIHSS score

SECONDARY OUTCOMES:
changed indication for surgery | 1 - 7 days before surgery
  towards surgery, avoids surgery towards biopsy, avoids surgery towards follow-up
change of the approach | 1 - 7 days before surgery
  using a different direct to approach the lesion (different sulcus, gyrus, sub cortically)
size of craniotomy | intraoperatively
  in mm ap and lateral
use of intraoperative motor mapping via MEP | intraoperatively
  yes/no
duration of intraoperative motor mapping via MEP | intraoperatively
  in min
duration of surgery | intraoperatively
  in min
extent of resection | intraoperatively
  in % via volumetry
use of further modalities (fMRI, DTI fiber tracking, SSEP phase reversal) | intraoperatively
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Sandro M Krieg, MD, MBA, Principal Investigator — Technical University of Munich
Locations (7):
- Germany (5):
  - Department of Neurosurgery, Klinikum rechts der Isar, TUM, Munich, Bavaria
  - Charité Universitätsmedizin Berlin, Berlin
  - Vivantes Klinikum Neu-Kölln, Berlin
  - Klinikum Bielefeld, Bielefeld
  - Klinikum Günzburg, Günzburg
- Department of Neurosurgery, University of Messina, Messina, Italy
- Universität Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No